CLINICAL TRIAL: NCT06014008
Title: The Effect of Lacticaseibacillus Paracasei Strain Shirota (LcS) in Healthy US Individuals Suffering From Hard or Lumpy Stools: A Randomized Controlled Open Trial.
Brief Title: Effect of L. Paracasei Strain Shirota on Constipation in Healthy US Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yakult U.S.A. Inc. (Industry)
Collaborators: BioFortis (Other); Dieta Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIO-2310
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Constipation
Keywords: probiotics; Lacticaseibacillus paracasei strain Shirota; Bristol stool form scale; imaging; constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention group (No Intervention): Not taking test product
- Test product consumption group (Experimental): Participants will take one bottle (80 ml) of Yakult® drink daily for a period of 4 weeks. Yakult is a branded probiotic drink with 8x10^9 CFU Lacticaseibacillus paracasei strain Shirota. Subsequently, a two-week follow-up period will follow.
  Interventions: Other: Test product consumption group

INTERVENTIONS:
Other: Test product consumption group — Participants will take one bottle (80 ml) of Yakult® drink daily for a period of 4 weeks. Yakult is a branded probiotic drink with 8x10^9 CFU Lacticaseibacillus paracasei strain Shirota. Subsequently, a two-week follow-up period will follow.
  Arms: Test product consumption group

SUMMARY:
The objective of this study is to investigate the efficacy of daily consumption of a fermented milk containing LcS in reducing the frequency of bowel movement with hard or lumpy stools in generally healthy U.S. adult population with intermittent bowel movements producing hard or lumpy stools.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 and <65 years old at Visit 1.
2. BMI between ≥18.5 to <30.0 kg/m2.
3. Has at least 3 bowel movements per week
4. ≥25% of bowel movements during the 2-week screening period produce hard or lumpy stools, defined as a Bristol Stool Form Scale (BSFS) score of 1 or 2 as determined from the participant's self-reported rating.
5. Regular breakfast consumer by self-report.
6. Has a smartphone supporting either iOS version 11.0 (or later) or Android version 5.0 (or later) operating software capable of downloading and running the Dieta Health app to collect study data.
7. Willing to consume the study product per the protocol instructions throughout the 28-day study intervention period.
8. Willing to maintain habitual dietary, lifestyle, and physical activity (with exceptions per study instructions) throughout the trial.
9. Willing to refrain from exclusionary medications, supplements, and products throughout the study.
10. Willing to limit alcohol consumption to ≤3 standard drinks/day and ≤7 standard drinks/week throughout the trial.
11. Non-user of tobacco or nicotine products or former user of any tobacco or nicotine product (not used within 6 months) and has no plans to change during the study period. Tobacco products include tobacco, smoking products (including, but not limited to cigarettes, cigars, chewing tobacco, e-cigarettes), and nicotine products (e.g., nicotine gum and/or nicotine patches) within 6 months of Visit 1 (Day 0) and during the study period.
12. Non-user or former user of any marijuana or hemp products (not used within 6 months) of Visit 1 (Day 0) and during the study period and has no plans to use marijuana or hemp products during the study period. No washout is required for topical marijuana or hemp products, but subjects are required to abstain from these products during the study period.
13. No health conditions that would prevent him/her from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history and screening physical exam.
14. Understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

1. Any known food allergies or intolerances to dairy or to any of the study product ingredients.
2. Consumption of probiotics or fermented products within 14 days of Visit 1 (Day 0) and during the study.
3. Presence of a clinically important GI condition that would potentially interfere with the evaluation of the study product (e.g., inflammatory bowel disease (IBD), irritable bowel syndrome (IBS), gastric reflux, indigestion, dyspepsia, Crohn's disease, celiac disease, history of surgery for weight loss, gastroparesis, and clinically significant lactose or gluten intolerance or other food or ingredient allergies). IBS will be determined as recurrent abdominal pain or discomfort at least 3 days/month in the last 3 months associated with: (a) improvement with defecation, (b) onset associated with change in frequency of stool, and (c) onset associated with a change in form (appearance of stool).
4. Constipation symptoms caused by primary organic disease of the colon or pelvic floor or, in the Investigator's opinion, caused by medication (e.g., morphine, codeine).
5. Uncontrolled and/or clinically important pulmonary (including uncontrolled asthma), hepatic, renal (except history of kidney stones in participants who are symptom free for 6 months), cardiac (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), endocrine (including Type 1 and Type 2 diabetes mellitus), hematologic, immunologic, neurologic (such as Alzheimer's or Parkinson's disease), psychiatric (including depression and/or anxiety disorders) or biliary condition(s). Conditions which are well-controlled or resolved will be assessed by the Clinical Investigator on a case-by-case basis.
6. Uncontrolled hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg) as defined by the blood pressure measured at Visit 1 (Day 0). Stable use of hypertension medication is allowed [defined as no change in medication regimen within 90 days of Visit 1 (Day 0)].
7. Weight loss or gain > 4.5 kg within 90 days of Visit 1 (Day 0), or currently or planning to be on a weight loss regimen or muscle-building/strengthening program during the study.
8. Signs or symptoms of an active infection of clinical relevance within 5 days of Visit 1 (Day 0). The visit may be rescheduled such that all signs and symptoms have resolved (at the discretion of the Clinical Investigator) at least 5 days prior to Visit 1 (Day 0).
9. Major trauma or any other surgical event within 90 days of Visit 1 (Day 0).
10. History or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
11. Use of proton pump inhibitors, H2 receptor antagonists, corticosteroids, antibiotics, antifungals, antiparasitics, antidiarrheals, and/or laxatives within 30 days of Visit 1 (Day 0).
12. Regular (>3 days/week) use of NSAIDs within 14 days of Visit 1 (Day 0).
13. Exposure to any non-registered drug product within 30 days prior to Visit 1 (Day 0).
14. Subject is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception during the study period. The method of contraception must be recorded.
15. Recent history (within 12 months of screening; Visit 1; Day 0) of alcohol or substance abuse. Alcohol abuse is defined as >14 drinks/week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
16. Recent (within 2 months) participation in any other clinical study prior to Visit 1 (Day 0).
17. Has a condition the Clinical Investigator believes would interfere with his/her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects that produce hard or lumpy stools (Subjectively evaluated Bristol stool form scale (BSFS) score of 1 or 2, ) ≥ 25% of bowel movements. | Four-week period from the start to the end of test product consumption.
  Compare the odds ratio of active to control of subjects with hard or lumpy stools (BSFS score of 1 or 2 as determined from the participant's self-reported rating) in at least 25% of the weekly bowel movements.

SECONDARY OUTCOMES:
Proportion of subjects that produce hard or lumpy stools (Objectively evaluated Bristol stool form scale (BSFS) score of 1 or 2, ) ≥ 25% of bowel movements. | Four-week period from the start to the end of test product consumption.
  Compare the odds ratio of active to control of subjects with hard or lumpy stools (BSFS score of 1 or 2 as determined by Dieta Health application stool image analysis) in at least 25% of the weekly bowel movements.
Odds ratio of active to control of subjects who had improved hard or lumpy stool ratio from baseline (BSFS score 1 or 2 as determined by Dieta Health application stool image analysis. | Four-week period from the start to the end of test product consumption.
Odds ratio of active to control of subjects who had improved hard or lumpy stool ratio from baseline (BSFS score 1 or 2 as determined from the participant's self-reported rating. | Four-week period from the start to the end of test product consumption.
Difference between groups in the stool consistency as collected by Dieta Health application stool image analysis. | Four-week period from the start to the end of test product consumption.
Difference between groups in the stool fuzziness as collected by Dieta Health application stool image analysis. | Four-week period from the start to the end of test product consumption.
Difference between groups in the stool fragmentation as collected by Dieta Health application stool image analysis. | Four-week period from the start to the end of test product consumption.
Difference between groups in the stool volume as collected by Dieta Health application stool image analysis. | Four-week period from the start to the end of test product consumption.
Difference between groups in the stool frequency as collected by Dieta Health application stool image analysis. | Four-week period from the start to the end of test product consumption.
Difference between groups in total and sub scores of PAC-QOL questionnaire. | Four-week period from the start to the end of test product consumption.
Difference between groups in the proportion of bowel movements having straining during evacuation. | Four-week period from the start to the end of test product consumption.
Difference between groups in the proportion of bowel movement having sensation of remaining stool in the rectum after evacuation. | Four-week period from the start to the end of test product consumption.

OTHER OUTCOMES:
Difference between groups in the Bristol stool form score of the first stool as collected by Dieta Health application stool image analysis after waking up. | Four-week period from the start to the end of test product consumption.
Difference between groups in the fuzziness of the first stool as collected by Dieta Health application stool image analysis after waking up. | Four-week period from the start to the end of test product consumption.
Difference between groups in the fragmentation of the first stool as collected by Dieta Health application stool image analysis after waking up. | Four-week period from the start to the end of test product consumption.
Difference between groups in the volume of the first stool as collected by Dieta Health application stool image analysis after waking up. | Four-week period from the start to the end of test product consumption.
Clustering analysis on the multivariate data and to identify distinct groups of subjects who receive benefit from the product. | Four-week period from the start to the end of test product consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Aditi Shah, MD, Principal Investigator — BioFortis
Locations (1):
- Biofortis, Chicago, Illinois, United States

REFERENCES:
- [Derived] Cook CM, Akiyama T, Blonquist T, Mah E, Derrig L, Shibata H. Effect of Daily Consumption of a Fermented Milk Containing Lacticaseibacillus paracasei Strain Shirota (LcS) on Stool Consistency in United States Adults with Hard or Lumpy Stools: A Randomized Controlled Trial. J Nutr. 2025 Apr;155(4):1183-1192. doi: 10.1016/j.tjnut.2025.02.021. Epub 2025 Feb 28. PMID 40024315